CLINICAL TRIAL: NCT00641056
Title: Efficacy of Once-Weekly Exenatide Long-Acting Release and Once-Daily Insulin Glargine in Patients With Type 2 Diabetes Treated With Metformin Alone or in Combination With Sulfonylurea
Brief Title: Efficacy of Exenatide Once Weekly and Once-Daily Insulin Glargine in Patients With Type 2 Diabetes Treated With Metformin Alone or in Combination With Sulfonylurea (DURATION - 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWBR (DURATION - 3)
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; exenatide once weekly; metformin; sulfonylurea; insulin glargine; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Exenatide Once Weekly
- 2 (Active Comparator)
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Exenatide Once Weekly — subcutaneous injection, 2.0mcg, once weekly
  Arms: 1
Drug: Insulin Glargine — subcutaneous injection, variable dose, QD
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of 2.0 mg exenatide once weekly and insulin glargine, titrated to glucose targets using the algorithm described by Yki- Järvinen et al.(2007), with respect to glycemic improvements, body weight, fasting lipids, safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes and at least 18 years of age at screening.
* Hemoglobin A1c (HbA1c) of 7.1% to 11.0%, inclusive, at screening.
* Body mass index (BMI) of 25 kg/m2 to 45 kg/m2, inclusive, at screening.
* Have a history of stable body weight (not varying by >5% for at least 3 months prior to screening).
* Have been treated with metformin(Met) for at least 3 months and have been taking a stable dose for at least 8 weeks prior to screening OR
* Have been treated with metformin(Met) for at least 3 months and have been taking a stable dose for at least 8 weeks prior to screening and have been treated with SU for at least 3 months and have been taking a stable dose of at least an optimally effective dose of brand of SU for 8 weeks prior to screening.

Exclusion Criteria:

* Have had a clinically significant history of cardiac disease or presence of active cardiac disease within the year prior to inclusion in the study, including myocardial infarction, clinically significant arrhythmia, unstable angina, moderate to severe congestive heart failure, coronary artery bypass surgery, or angioplasty; or is expected to require coronary artery bypass surgery or angioplasty during the course of the study.
* Have clinical signs or symptoms of liver disease, acute or chronic hepatitis.
* Have a history of renal transplantation or are currently receiving renal dialysis.
* Have active or untreated malignancy, or have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have had greater than three episodes of major hypoglycemia within 6 months prior to screening.
* Have any contraindication for the oral antidiabetic agent which they use.
* Have a known allergy or hypersensitivity to insulin glargine, exenatide once weekly, or excipients contained in these agents.
* Are known to have active proliferative retinopathy.
* Have been treated with drugs that promote weight loss (e.g., Xenical® [orlistat], Meridia® [sibutramine], Acomplia® [rimonabant], Acutrim® [phenylpropanolamine], or similar over-the-counter medications) within 3 months of screening.
* Have been treated for longer than 2 weeks with any of the following excluded medications within 3 months prior to screening:

  * Insulin
  * Thiazolidinediones (e.g., Actos® [pioglitazone] or Avandia® [rosiglitazone])
  * Alpha-glucosidase inhibitors (e.g., Glyset® [miglitol] or Precose® [acarbose])
  * Meglitinides (e.g., Prandin® [repaglinide] or Starlix® [nateglinide]).
  * Byetta® (exenatide BID formulation)
  * Dipeptidyl peptidase (DPP)-4 inhibitors (e.g., Januvia™ [sitagliptin], Galvus® [vildagliptin])
  * Symlin® (pramlintide acetate).
* Have had an organ transplant.
* Have donated blood within 30 days of screening.
* Have previously completed or withdrawn from this study or any other study investigating exenatide once weekly.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Are currently enrolled in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (75):
- United States (12):
  - Research Site, Escondido, California
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Idaho Falls, Idaho
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Dayton, Ohio
  - Research Site, Ada, Oklahoma
  - Research Site, San Antonio, Texas
  - Research Site, Spokane, Washington
- Australia (6):
  - Research Site, Wollongong, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Keswick, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Geelong, Victoria
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Edegem
- Czechia (3):
  - Research Site, Mělník
  - Research Site, Prague
  - Research Site, Stodůlky
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Arhus C
  - Research Site, Herlev
  - Research Site, Køge
- France (5):
  - Research Site, Angers
  - Research Site, Corbeil Essoness
  - Research Site, Nancy
  - Research Site, Nanterre
  - Research Site, Toulouse
- Germany (9):
  - Research Site, Bad Mergentheim
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Falkensee
  - Research Site, Fulda
  - Research Site, Münster
  - Research Site, Othmarschen
  - Research Site, Rothenburg An Der Fulda
  - Research Site, Speyer
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Pécs
- Mexico (4):
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, Tampico
  - Research Site, Tijuana
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Gouda
  - Research Site, Hoogeveen
  - Research Site, Rotterdam
  - Research Site, Zwijndrecht
  - Research Site, Zwolle
- Puerto Rico (2):
  - Research Site, Caguas
  - Research Site, Yabucoa
- Russia (3):
  - Research Site, Moscow
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (7):
  - Research Site, Alicante
  - Research Site, Alzira-Valencia
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Teruel
- Taiwan (4):
  - Research Site, Chiayi City
  - Research Site, Tainan County
  - Research Site, Taipei
  - Research Site, Taoyuan District

REFERENCES:
- [Result] Diamant M, Van Gaal L, Stranks S, Guerci B, MacConell L, Haber H, Scism-Bacon J, Trautmann M. Safety and efficacy of once-weekly exenatide compared with insulin glargine titrated to target in patients with type 2 diabetes over 84 weeks. Diabetes Care. 2012 Apr;35(4):683-9. doi: 10.2337/dc11-1233. Epub 2012 Feb 22. PMID 22357185
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296
- [Derived] Diamant M, Van Gaal L, Guerci B, Stranks S, Han J, Malloy J, Boardman MK, Trautmann ME. Exenatide once weekly versus insulin glargine for type 2 diabetes (DURATION-3): 3-year results of an open-label randomised trial. Lancet Diabetes Endocrinol. 2014 Jun;2(6):464-73. doi: 10.1016/S2213-8587(14)70029-4. Epub 2014 Apr 4. PMID 24731672
- [Derived] Grimm M, Han J, Weaver C, Griffin P, Schulteis CT, Dong H, Malloy J. Efficacy, safety, and tolerability of exenatide once weekly in patients with type 2 diabetes mellitus: an integrated analysis of the DURATION trials. Postgrad Med. 2013 May;125(3):47-57. doi: 10.3810/pgm.2013.05.2660. PMID 23748506
- [Derived] Meloni AR, DeYoung MB, Han J, Best JH, Grimm M. Treatment of patients with type 2 diabetes with exenatide once weekly versus oral glucose-lowering medications or insulin glargine: achievement of glycemic and cardiovascular goals. Cardiovasc Diabetol. 2013 Mar 23;12:48. doi: 10.1186/1475-2840-12-48. PMID 23522121
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] Diamant M, Van Gaal L, Stranks S, Northrup J, Cao D, Taylor K, Trautmann M. Once weekly exenatide compared with insulin glargine titrated to target in patients with type 2 diabetes (DURATION-3): an open-label randomised trial. Lancet. 2010 Jun 26;375(9733):2234-43. doi: 10.1016/S0140-6736(10)60406-0. PMID 20609969

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly: Patients assigned to the Exenatide Once Weekly group received a 2 mg dose of exenatide injected once a week.
- Insulin Glargine: Patients assigned to the Insulin Glargine group started insulin glargine treatment with 10 units per day, utilizing the INITIATE (Initiate Insulin by Aggressive Titration and Education) dosing and were instructed to adjust insulin doses to achieve a target blood glucose of 4.0-5.5 mmol/L.
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Started | 233 | 234
Intent to Treat (ITT) | 233 | 223
Completed | 204 | 209
Not Completed | 29 | 25
Not completed — Adverse Event | 12 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Entry Criteria Not Met | 3 | 0
Not completed — Subject Decision | 6 | 19
Not completed — Sponsor Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Insulin Glargine | Total
Number analyzed (Participants) | 233 | 223 | 456
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 184 | 167 | 351
  >=65 years | 49 | 56 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.72) | 58.3 (9.08) | 57.9 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 100 | 213
  Male | 120 | 123 | 243
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.32 (1.094) | 8.29 (1.020) | 8.31 (1.057)
Weight [Mean (Standard Deviation); unit: kg] | 91.22 (18.582) | 90.56 (16.348) | 90.90 (17.509)
Background Oral Antidiabetic Agent (OAD) [Number; unit: participants]
  Metformin (Met) | 164 | 157 | 321
  Met+Sulfonylurea (SU) | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Change in HbA1c from baseline to Week 26
Time Frame: Baseline, Week 26
Population: ITT Population: All randomized patients who had taken at least one dose of study drug. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 205 | 206
percentage of total hemoglobin | -1.47 (0.05) | -1.31 (0.06)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Mixed-model Repeated Measures (MMRM) Analysis of Covariance (ANCOVA) model includes treatment, baseline HbA1c, country, background OAD stratum, week of visit, and treatment-by-week interaction as fixed effects; patient and error as random effects. Superiority of exenatide once weekly to insulin glargine is concluded if the upper limit of the 95% confidence interval for the treatment difference [exenatide once weekly-insulin glargine]<0; noninferiority is concluded if this upper limit<0.3%; Test type: Non-Inferiority or Equivalence — Power: 205 patients per treatment group would provide approximately 92% power to detect a true difference between treatments of 0.4% in change in HbA1c from baseline with a 2-sided t test at a significance level of 0.05, assuming a common standard deviation of 1.2%; p = 0.017, Mixed Models Analysis — No adjustments for multiplicity were performed; Least Squares Mean Difference = -0.16, 95% CI 2-sided [-0.29 to -0.03], Standard Error of Mean 0.07

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <=7.0% at Week 26
Description: Percentage of patients achieving HbA1c <=7.0% at Week 26 (for patients with HbA1c >7% at baseline)
Time Frame: Baseline, Week 26
Population: ITT Population. Only patients with baseline HbA1c > 7% were included in calculation. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 209 | 207
percentage of patients | 62.2 | 54.1
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Percentage of patients achieving HbA1c <=7.0% at Week 26 were compared between treatments using a Cochran-Mantel-Haenszel (CMH) test, in which background OAD and country served as the stratification factors; Test type: Superiority or Other; p = 0.097, Cochran-Mantel-Haenszel — No adjustments for multiplicity were performed

3. Secondary Outcome: Percentage of Patients Achieving HbA1c <=6.5% at Week 26
Description: Percentage of patients achieving HbA1c <=6.5% at Week 26 (for patients with HbA1c >6.5% at baseline)
Time Frame: Baseline, Week 26
Population: ITT Population. Only patients with baseline HbA1c > 6.5% were included in calculation. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 227 | 218
percentage of patients | 43.2 | 28.4
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Percentage of patients achieving HbA1c <=6.5% at Week 26 were compared between treatments using a CMH test, in which background OAD and country served as the stratification factors; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — No adjustments for multiplicity were performed

4. Secondary Outcome: Change in Fasting Serum Glucose (FSG) From Baseline to Week 26
Description: Change in FSG (mmol/L) from Baseline to Week 26
Time Frame: Baseline, Week 26
Population: ITT Population. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 192 | 197
mmol/L | -2.13 (0.16) | -2.76 (0.16)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; MMRM ANCOVA with change in FSG as the dependent variable; treatment, baseline FSG, country, background OAD stratum, week of visit, and treatment-by-week interaction as fixed effects; patient and error as random effects; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — No adjustments for multiplicity were performed; Least Squares Mean Difference = 0.63, 95% CI 2-sided [0.25 to 1.00], Standard Error of Mean 0.19

5. Secondary Outcome: Change in Body Weight (BW) From Baseline to Week 26
Description: Change in BW (kg) from Baseline to Week 26
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 207 | 209
kg | -2.63 (0.20) | 1.42 (0.20)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; MMRM ANCOVA with change in BW as the dependent variable; treatment, baseline BW, country, background OAD stratum, week of visit, and treatment-by-week interaction as fixed effects; patient and error as random effects; Test type: Superiority or Other; p < .001, Mixed Models Analysis — No adjustments for multiplicity were performed; Least Squares Mean Difference = -4.05, 95% CI 2-sided [-4.57 to -3.52], Standard Error of Mean 0.27

6. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 26
Description: Change in Total Cholesterol (mmol/L) from Baseline to Week 26
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 191 | 198
mmol/L | -0.12 (0.06) | -0.04 (0.06)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; MMRM ANCOVA with change in total cholesterol as the dependent variable; treatment, baseline total cholesterol, country, background OAD stratum, week of visit, and treatment-by-week interaction as fixed effects; patient and error as random effects; Test type: Superiority or Other; p = 0.292, Mixed Models Analysis — No adjustments for multiplicity were performed; Least Squares Mean Difference = -0.07, 95% CI 2-sided [-0.21 to 0.06], Standard Error of Mean 0.07

7. Secondary Outcome: Change in High-density Lipoprotein Cholesterol (HDL) From Baseline to Week 26
Description: Change in HDL (mmol/L) from Baseline to Week 26
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 191 | 198
mmol/L | -0.00 (0.01) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; MMRM ANCOVA with change in HDL as the dependent variable; treatment, baseline HDL, country, background OAD stratum, week of visit, and treatment-by-week interaction as fixed effects; patient and error as random effects; Test type: Superiority or Other; p = 0.377, Mixed Models Analysis — No adjustments for multiplicity were performed; Least Squares Mean Difference = -0.02, 95% CI 2-sided [-0.05 to 0.02], Standard Error of Mean 0.02

8. Secondary Outcome: Ratio of Triglycerides at Week 26 to Baseline
Description: Ratio of Triglycerides (measured in mmol/L) at Week 26 to Baseline. Log (Postbaseline Triglycerides) - log (Baseline Triglycerides); change from baseline to endpoint is presented as ratio of endpoint to baseline.
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 191 | 198
ratio | 0.96 (0.03) | 0.89 (0.03)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Triglycerides data were logarithm-transformed and the change at Week 26 to baseline, expressed as the ratio, was analyzed by MMRM ANCOVA with change in triglycerides as the dependent variable; treatment, baseline triglycerides, country, background OAD stratum, week of visit, and treatment-by-week interaction as fixed effects; patient and error as random effects; Test type: Superiority or Other; p = 0.077, Mixed Models Analysis — No adjustments for multiplicity were performed; Geometric Least Squares Mean Ratio = 1.07, 95% CI 2-sided [0.99 to 1.15], Standard Error of Mean 0.04

9. Secondary Outcome: Change in Blood Pressure From Baseline to Week 26
Description: Change in Systolic Blood Pressure (mmHg) and Diastolic Blood Pressure (mmHg) from Baseline to Week 26
Time Frame: Baseline, Week 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 233 | 222
mmHg
  Systolic Blood Pressure | -3.03 (16.57) | -0.63 (14.88)
  Diastolic Blood Pressure | -1.15 (10.08) | -0.72 (8.73)

10. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Hypoglycemic Episodes
Description: Major hypoglycemia: any episode with symptoms consistent with hypoglycemia that resulted in loss of consciousness or seizure with prompt recovery in response to administration of glucagon or glucose or documented hypoglycemia (blood glucose <3.0 mmol/L [54 mg/dL]) and required the assistance of another person. Minor hypoglycemia: any time a patient felt that he or she was experiencing a sign or symptom of hypoglycemia that was self-treated or resolved on its own and had a blood glucose level <3.0 mmol/L (54 mg/dL) and not classified as major hypoglycemia.
Time Frame: Baseline to Week 26
Population: ITT Population.
Measure: Mean (Standard Error); unit: rate per subject-year
Groups:
- Exenatide Once Weekly With SU: Patients assigned to the Exenatide Once Weekly With SU group received a 2 mg dose of exenatide injected once a week and took concomitant Met+SU.
- Insulin Glargine With SU: Patients assigned to the Insulin Glargine with SU group started insulin glargine treatment with 10 units per day, utilizing the INITIATE (Initiate Insulin by Aggressive Titration and Education) dosing and were instructed to adjust insulin doses to achieve a target blood glucose of 4.0-5.5 mmol/L and took concomitant Met+SU.
- Exenatide Once Weekly No SU: Patients assigned to the Exenatide Once Weekly No SU group received a 2 mg dose of exenatide injected once a week and took concomitant Met only.
- Insulin Glargine No SU: Patients assigned to the Insulin Glargine No SU group started insulin glargine treatment with 10 units per day, utilizing the INITIATE (Initiate Insulin by Aggressive Titration and Education) dosing and were instructed to adjust insulin doses to achieve a target blood glucose of 4.0-5.5 mmol/L and took concomitant Met only.
Arm/Group | Exenatide Once Weekly With SU | Insulin Glargine With SU | Exenatide Once Weekly No SU | Insulin Glargine No SU
Number analyzed (Participants) | 69 | 66 | 164 | 157
rate per subject-year
  Major Hypoglycemia | 0.00 (0.000) | 0.03 (0.030) | 0.01 (0.013) | 0.01 (0.013)
  Minor Hypoglycemia | 1.14 (0.184) | 2.66 (0.284) | 0.10 (0.037) | 0.63 (0.091)

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 11/233 | 10/223
Other Adverse Events (participants affected / at risk) | 100/233 | 52/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=233) | Insulin Glargine (N=223)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardioversion (Surgical and medical procedures) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Injection site nodule (General disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral pericarditis (Infections and infestations) | 1 | 0
Vitrectomy (Surgical and medical procedures) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Colon polypectomy (Surgical and medical procedures) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Peripheral nerve transposition (Surgical and medical procedures) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=233) | Insulin Glargine (N=223)
Nasopharyngitis (Infections and infestations) | 30 | 39
Nausea (Gastrointestinal disorders) | 30 | 3
Headache (Nervous system disorders) | 23 | 16
Diarrhoea (Gastrointestinal disorders) | 20 | 8
Injection site nodule (General disorders) | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days